CLINICAL TRIAL: NCT00701103
Title: An Open-Label, Dose Escalation Phase I Trial of MK-0646 Given as a Once Weekly, Every Other Week, or Every Three Week Infusion in Patients With Advanced Solid Tumors and Multiple Myeloma
Brief Title: Dose Escalation Trial of Dalotuzumab (MK-0646) in Advanced Solid Tumors and Multiple Myeloma (MK-0646-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0646-001; 2007_660 (Other: Merck Telerex Number); NCT00282737 (obsolete NCT alias)
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Solid Tumor; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — dalotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- Dalotuzumab 1.25 mg/kg Q1W (10 mg/mL) (Experimental): Participants received dalotuzumab 1.25 mg/kg (10 mg/mL) intravenous (IV) infusion 1 time every 1 week (Q1W).
  Interventions: Drug: Dalotuzumab
- Dalotuzumab 2.5 mg/kg Q1W (10 mg/mL) (Experimental): Participants received dalotuzumab 2.5 mg/kg (10 mg/mL) IV infusion Q1W.
  Interventions: Drug: Dalotuzumab
- Dalotuzumab 5 mg/kg Q1W (10 mg/mL) (Experimental): Participants received dalotuzumab 5 mg/kg (10 mg/mL) IV infusion Q1W.
  Interventions: Drug: Dalotuzumab
- Dalotuzumab 10 mg/kg Q1W (10 mg/mL) (Experimental): Participants received dalotuzumab 10 mg/kg (10 mg/mL) IV infusion Q1W.
  Interventions: Drug: Dalotuzumab
- Dalotuzumab 10 mg/kg Q1W (20 mg/mL) (Experimental): Participants received dalotuzumab 10 mg/kg (20 mg/mL) IV infusion Q1W.
  Interventions: Drug: Dalotuzumab
- Dalotuzumab 15 mg/kg Q1W (10 mg/mL) (Experimental): Participants received dalotuzumab 15 mg/kg (10 mg/mL) IV infusion Q1W.
  Interventions: Drug: Dalotuzumab
- Dalotuzumab 15 mg/kg Q1W (20 mg/mL) (Experimental): Participants received dalotuzumab 15 mg/kg (20 mg/ mL) IV infusion Q1W.
  Interventions: Drug: Dalotuzumab
- Dalotuzumab 20 mg/kg Q1W (10 mg/mL) (Experimental): Participants received dalotuzumab 20 mg/kg (10 mg/mL) IV infusion Q1W.
  Interventions: Drug: Dalotuzumab
- Dalotuzumab 20 mg/kg Q1W (20 mg/mL) (Experimental): Participants received dalotuzumab 20.0 mg/kg (20 mg/mL) IV infusion Q1W.
  Interventions: Drug: Dalotuzumab
- Dalotuzumab 20 mg/kg Q2W (20 mg/mL) (Experimental): Participants received dalotuzumab 20 mg/kg (20 mg/mL) IV infusion 1 time every 2 weeks (Q2W).
  Interventions: Drug: Dalotuzumab
- Dalotuzumab 30 mg/kg Q3W (20 mg/mL) (Experimental): Participants received dalotuzumab 30 mg/kg (20 mg/mL) IV infusion1 time every 3 weeks (Q3W).
  Interventions: Drug: Dalotuzumab

INTERVENTIONS:
Drug: Dalotuzumab — IV infusion
  Other Names: MK-0646

SUMMARY:
This study will look for the highest tolerated dose of dalotuzumab (MK-0646) given as weekly, every other week. or a every three week infusion.

The hypothesis of this study is that administration of dalotuzumab as a one- to two-hour weekly, every other week, or every three week infusion in participants with advanced cancer will be generally safe and tolerated at a dose which achieves a trough concentration ≥3 μg/mL.

DETAILED DESCRIPTION:
Trial Duration of Treatment: Participants can be treated for up to two years if their disease has not progressed and they are not having unmanageable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Participant has metastatic or locally advanced solid tumor or multiple myeloma
* Tumor specimen has IGF-1R expression
* Participant agrees to use birth control throughout study

Exclusion Criteria:

* Participant must not be recovering from antineoplastic therapy in the last 4 weeks
* Participant has participated in a clinical trial in the last 4 weeks
* Participant has a history of heart problems such as congestive heart failure, angina, heart attack or stroke in the last 3 months
* Participant is taking growth hormone or growth hormone inhibitors
* If female, participant is pregnant or breastfeeding
* Participant is human immunodeficiency virus (HIV) positive
* Participant has a history of hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-01-12 (Actual); Primary Completion 2009-12-01 (Actual); Study Completion 2009-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Atzori F, Tabernero J, Cervantes A, Prudkin L, Andreu J, Rodriguez-Braun E, Domingo A, Guijarro J, Gamez C, Rodon J, Di Cosimo S, Brown H, Clark J, Hardwick JS, Beckman RA, Hanley WD, Hsu K, Calvo E, Rosello S, Langdon RB, Baselga J. A phase I pharmacokinetic and pharmacodynamic study of dalotuzumab (MK-0646), an anti-insulin-like growth factor-1 receptor monoclonal antibody, in patients with advanced solid tumors. Clin Cancer Res. 2011 Oct 1;17(19):6304-12. doi: 10.1158/1078-0432.CCR-10-3336. Epub 2011 Aug 2. PMID 21810918

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were ≥18 years old, had metastatic or locally advanced solid tumors (including multiple myeloma) and failed to respond to standard therapy, or had progressed despite standard therapy, or for whom standard therapy did not exist were recruited for this study.
Groups:
- Dalotuzumab 30 mg/kg Q3W (20 mg/mL): Participants received dalotuzumab 30 mg/kg (20 mg/mL) IV infusion 1 time every 3 weeks (Q3W).
Period: Overall Study
Arm/Group | Dalotuzumab 1.25 mg/kg Q1W (10 mg/mL) | Dalotuzumab 2.5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (20 mg/mL) | Dalotuzumab 15 mg/kg Q1W (10 mg/mL) | Dalotuzumab 15 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q1W (10 mg/mL) | Dalotuzumab 20 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q2W (20 mg/mL) | Dalotuzumab 30 mg/kg Q3W (20 mg/mL)
Started | 5 | 3 | 8 | 6 | 6 | 6 | 8 | 7 | 9 | 11 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 3 | 8 | 6 | 6 | 6 | 8 | 7 | 9 | 11 | 11
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Not completed — Progressive Disease | 5 | 2 | 6 | 5 | 6 | 5 | 7 | 7 | 8 | 8 | 11
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The population consisted of all participants who received at least one dose of study drug.
Groups:
- Dalotuzumab 1.25 mg/kg Q1W (10 mg/mL): Participants received dalotuzumab 1.25 mg/kg (10 mg/mL) IV infusion Q1W.
- Dalotuzumab 20 mg/kg Q2W (20 mg/mL): Participants received dalotuzumab 20 mg/kg (20 mg/mL) IV infusion Q2W.
- Dalotuzumab 30 mg/kg Q3W (20 mg/mL): Participants received dalotuzumab 30 mg/kg (20 mg/mL) IV infusion Q3W.
- Total: Total of all reporting groups
Arm/Group | Dalotuzumab 1.25 mg/kg Q1W (10 mg/mL) | Dalotuzumab 2.5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (20 mg/mL) | Dalotuzumab 15 mg/kg Q1W (10 mg/mL) | Dalotuzumab 15 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q1W (10 mg/mL) | Dalotuzumab 20 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q2W (20 mg/mL) | Dalotuzumab 30 mg/kg Q3W (20 mg/mL) | Total
Number analyzed (Participants) | 5 | 3 | 8 | 6 | 6 | 6 | 8 | 7 | 9 | 11 | 11 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69 (9) [59 to 81] | 60 (9) [50 to 68] | 68 (9) [51 to 80] | 56 (10) [40 to 68] | 53 (17) [26 to 70] | 49 (22) [23 to 70] | 54 (18) [29 to 64] | 46 (13) [27 to 78] | 52 (18) [22 to 69] | 55 (17) [23 to 77] | 52 (15) [19 to 73] | 55 (16) [19 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 4 | 6 | 3 | 3 | 4 | 2 | 5 | 5 | 6 | 40
  Male | 4 | 2 | 4 | 0 | 3 | 3 | 4 | 5 | 4 | 6 | 5 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced One or More Dose-limiting Toxicities (DLTs)
Description: Toxicity was graded and recorded according to National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events version 3.0 (CTCAE 3.0). A DLT was defined as any Grade 3 or 4 toxicity. A Grade 3 toxicity was defined as severe or medically significant but not immediately life-threatening OR hospitalization or prolongation of hospitalization indicated OR disabling OR limiting self care activities of daily living. A Grade 4 toxicity was defined as: life-threatening consequences OR urgent intervention indicated. Participants were monitored for the occurrence of DLTs during the first 3 weeks of dosing with dalotuzumab.
Time Frame: Up to 3 weeks
Population: The population consisted of all participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dalotuzumab 1.25 mg/kg Q1W (10 mg/mL) | Dalotuzumab 2.5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (20 mg/mL) | Dalotuzumab 15 mg/kg Q1W (10 mg/mL) | Dalotuzumab 15 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q1W (10 mg/mL) | Dalotuzumab 20 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q2W (20 mg/mL) | Dalotuzumab 30 mg/kg Q3W (20 mg/mL)
Number analyzed (Participants) | 5 | 3 | 8 | 6 | 6 | 6 | 8 | 7 | 9 | 11 | 11
Percentage of Participants | 0 | 0 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Mean Terminal Half-life (t1/2) of Dalotuzumab
Description: Terminal half-life is defined as the time it takes for the blood plasma concentration of a substance to halve (plasma half-life). Blood samples for measurement of serum levels of dalotuzumab were obtained at: pre-dose; pre-end infusion; 0.5, 5, 10, 24, 30 (Q1W only), 48, 96, 168 (Q2W/Q3W only), 336 (Q3W only) hours post infusion. For infusions >1 hour in duration, an additional sample was obtained at the mid-point of the infusion. Data presented are for the harmonic mean t1/2 for dalotuzumab.
Time Frame: Predose; pre-end infusion; 0.5, 5, 10, 24, 30 (Q1W only), 48, 96, 168 (Q2W/Q3W only), 336 (Q3W only) hours post-infusion
Population: The population consisted of all evaluable participants who received >90% of intended drug volume and had t1/2 pharmacokinetic measurements at Baseline and at least once during treatment.
Measure: Mean (Full Range); unit: Hours
Arm/Group | Dalotuzumab 1.25 mg/kg Q1W (10 mg/mL) | Dalotuzumab 2.5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (20 mg/mL) | Dalotuzumab 15 mg/kg Q1W (10 mg/mL) | Dalotuzumab 15 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q1W (10 mg/mL) | Dalotuzumab 20 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q2W (20 mg/mL) | Dalotuzumab 30 mg/kg Q3W (20 mg/mL)
Number analyzed (Participants) | 5 | 3 | 8 | 6 | 3 | 6 | 8 | 7 | 9 | 11 | 11
Hours | 67 [46 to 121] | 79 [53 to 113] | 83 [41 to 240] | 169 [134 to 265] | 100 [81 to 123] | 95 [43 to 165] | 110 [83 to 215] | 129 [74 to 240] | 120 [66 to 184] | 106 [44 to 134] | 142 [73 to 187]

3. Primary Outcome: Area Under the Time-concentration Curve From 0 to Infinity Hours (AUC0-∞) of Dalotuzumab
Description: AUC0-∞ represents the total drug exposure over time. Blood samples for measurement of serum levels of dalotuzumab were obtained at: Predose; pre-end infusion; 0.5, 5, 10, 24, 30 (Q1W only), 48, 96, 168 (Q2W/Q3W only), 336 (Q3W only) hours post-infusion. For infusions >1 hour in duration, an additional sample was obtained at the mid-point of the infusion.
Time Frame: as for outcome 2
Population: The population consisted of all evaluable participants who received >90% of intended drug volume and had AUC0-last pharmacokinetic measurements at Baseline and at least once during treatment.
Measure: Mean (Standard Deviation); unit: mg*hr/mL
Arm/Group | Dalotuzumab 1.25 mg/kg Q1W (10 mg/mL) | Dalotuzumab 2.5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (20 mg/mL) | Dalotuzumab 15 mg/kg Q1W (10 mg/mL) | Dalotuzumab 15 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q1W (10 mg/mL) | Dalotuzumab 20 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q2W (20 mg/mL) | Dalotuzumab 30 mg/kg Q3W (20 mg/mL)
Number analyzed (Participants) | 5 | 3 | 8 | 6 | 3 | 6 | 8 | 7 | 9 | 11 | 11
mg*hr/mL | 1.6 (0.4) | 3.7 (1.1) | 12.9 (4.4) | 28.9 (10.4) | 18.4 (4.1) | 39.4 (14.5) | 28.8 (8.8) | 52.7 (19.2) | 44.3 (20.0) | 45.9 (14.4) | 92.6 (29.8)

4. Primary Outcome: Mean Serum Clearance of Dalotuzumab
Description: Clearance is defined as the volume of serum from which study drug was completely removed per unit of time. Blood samples for measurement of serum levels of dalotuzumab were obtained at: pre-dose; pre-end infusion; 0.5, 5, 10, 24, 30 (Q1W only), 48, 96, 168 (Q2W/Q3W only), 336 (Q3W only) hours post infusion. For infusions >1 hour in duration, an additional sample was obtained at the mid-point of the infusion.
Time Frame: as for outcome 2
Population: The population consisted of all evaluable participants who received >90% of intended drug volume and had mean serum clearance pharmacokinetic measurements at Baseline and at least once during treatment.
Measure: Mean (Standard Deviation); unit: mL/min/kg
Arm/Group | Dalotuzumab 1.25 mg/kg Q1W (10 mg/mL) | Dalotuzumab 2.5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (20 mg/mL) | Dalotuzumab 15 mg/kg Q1W (10 mg/mL) | Dalotuzumab 15 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q1W (10 mg/mL) | Dalotuzumab 20 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q2W (20 mg/mL) | Dalotuzumab 30 mg/kg Q3W (20 mg/mL)
Number analyzed (Participants) | 5 | 3 | 8 | 6 | 3 | 6 | 8 | 7 | 9 | 11 | 11
mL/min/kg | 0.013 (0.004) | 0.012 (0.003) | 0.007 (0.003) | 0.006 (0.002) | 0.009 (0.002) | 0.007 (0.004) | 0.010 (0.004) | 0.007 (0.003) | 0.009 (0.004) | 0.008 (0.003) | 0.006 (0.003)

5. Primary Outcome: Mean Trough Serum Concentration (Ctrough) of Dalotuzumab
Description: The lowest (trough) concentration of dalotuzumab prior to the next dose of dalotuzumab was measured.
Time Frame: Pre-dose immediately prior to second infusion: 168 hours for Q1W, 336 hours for Q2W and 504 hours for Q3W dosing
Population: The population consisted of all evaluable participants who received >90% of intended drug volume and had mean trough serum concentration pharmacokinetic measurements at Baseline and at least once during treatment.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Dalotuzumab 1.25 mg/kg Q1W (10 mg/mL) | Dalotuzumab 2.5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (20 mg/mL) | Dalotuzumab 15 mg/kg Q1W (10 mg/mL) | Dalotuzumab 15 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q1W (10 mg/mL) | Dalotuzumab 20 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q2W (20 mg/mL) | Dalotuzumab 30 mg/kg Q3W (20 mg/mL)
Number analyzed (Participants) | 5 | 3 | 8 | 6 | 3 | 6 | 8 | 7 | 9 | 11 | 11
ug/mL | 2.4 (2.2) | 7.2 (3.0) | 21.2 (8.3) | 54.8 (13.3) | 45.2 (17.4) | 81.2 (38.6) | 59.6 (17.3) | 110.5 (46.0) | 87.3 (41.5) | 57.0 (22.7) | 70.4 (34.1)

6. Secondary Outcome: Change From Baseline in Insulin-like Growth Factor Receptor Type 1 (IGF-1R) Protein Expression Level H-score in Skin Samples
Description: IGF-1R expression was measured in pre- and post-dose skin biopsy samples using an immunohistochemistry (IHC) assay as a function of time and dose. Results were expressed as an IGF-1R membrane H-score which could range from 0 to 300; with a score of 0 representing the absence of IGF-1R expression and an H-score of 300 representing maximum IGF-1R expression. Changes in IGF-1R expression levels from Baseline are summarized for all participants for whom these paired data were available. A post-dose decrease in IGF-1R membrane H-score was an indication of target engagement by dalotuzumab. A larger decrease in H-score correlated with a greater target engagement.
Time Frame: Predose in Cycle 1 (Baseline) and predose in Cycle 3 (Week 4)
Population: The population consisted of all evaluable participants who received >90% of intended drug volume and had skin IGF-1R pharmacodynamics measurements at Baseline and at least once during treatment. No data were available for the Dalotuzumab 30 mg/kg Q3W treatment group.
Measure: Mean (Standard Deviation); unit: H-score
Groups:
- Dalotuzumab 10 mg/kg Q1W (10 mg/mL): Participants received dalotuzumab 10 mg/kg IV infusion Q1W.
- Dalotuzumab 15 mg/kg Q1W (10 mg/mL): Participants received dalotuzumab 15 mg/kg IV infusion Q1W.
- Dalotuzumab 20 mg/kg Q1W (10 mg/mL): Participants received dalotuzumab 20 mg/kg IV infusion Q1W or Q2W.
Arm/Group | Dalotuzumab 1.25 mg/kg Q1W (10 mg/mL) | Dalotuzumab 2.5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (10 mg/mL) | Dalotuzumab 15 mg/kg Q1W (10 mg/mL) | Dalotuzumab 20 mg/kg Q1W (10 mg/mL) | Dalotuzumab 30 mg/kg Q3W (20 mg/mL)
Number analyzed (Participants) | 3 | 3 | 7 | 11 | 10 | 15 | 0
H-score
  Baseline | 186.7 (35.1) | 203.3 (55.1) | 218.6 (57.9) | 171.8 (40.2) | 182.0 (33.9) | 146.3 (76.9) |
  Change from Baseline | -1.7 (42.5) | -11.7 (48.6) | -20.0 (68.6) | -2.7 (42.2) | -39.0 (36.3) | -27.0 (54.1) |

7. Secondary Outcome: Change From Baseline in IGF-1R Protein Expression Level H-score in Tumor Samples
Description: IGF-1R expression was measured in pre- and post-dose tumor biopsy samples using an IHC assay as a function of time and dose. Results were expressed as an IGF-1R membrane H-score which could range from 0 to 300; with a score of 0 representing the absence of IGF-1R expression and an H-score of 300 representing maximum IGF-1R expression. Changes in IGF-1R expression levels from Baseline are summarized for all participants for whom these paired data were available. A post-dose decrease in IGF-1R membrane H-score was an indication of target engagement by dalotuzumab. A larger decrease in H-score correlated with a greater target engagement.
Time Frame: Predose in Cycle 1 (Baseline) and predose in Cycle 3 (Week 4)
Population: The population consisted of all evaluable participants who received >90% of intended drug volume and had IGF-1R tumor pharmacodynamics measurements at Baseline and at least once during treatment. No data were available for the Dalotuzumab 2.5 mg/kg Q1W and Dalotuzumab 30 mg/kg Q3W treatment groups.
Measure: Mean (Standard Deviation); unit: H-score
Arm/Group | Dalotuzumab 1.25 mg/kg Q1W (10 mg/mL) | Dalotuzumab 2.5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (10 mg/mL) | Dalotuzumab 15 mg/kg Q1W (10 mg/mL) | Dalotuzumab 20 mg/kg Q1W (10 mg/mL) | Dalotuzumab 30 mg/kg Q3W (20 mg/mL)
Number analyzed (Participants) | 2 | 0 | 5 | 4 | 7 | 15 | 0
H-score
  Baseline | 145.0 (91.9) |  | 84.0 (59.0) | 110.0 (46.9) | 134.3 (77.0) | 152.5 (72.4) |
  Change from Baseline | -80.0 (28.3) |  | -16.0 (27.0) | 10.0 (76.2) | -30.0 (40.0) | -40.8 (108.1) |

8. Secondary Outcome: Percentage of Participants Who Developed a Serum Human-anti-humanized-antibody (HAHA) Response to Dalotuzumab
Description: It is thought that the formation of HAHAs may block efficacy by prematurely clearing dalotuzumab and limit the possibility of future dalotuzumab therapy. Blood samples for the measurement of serum levels of HAHAs were obtained prior to treatment with dalotuzumab, and pre-dose Week 2 (Q1W), pre-dose Week 3 (Q2W), pre-dose Week 4 (QW3), pre-dose Week 5 (Q1W/Q2W), pre-dose Week 7 (Q2W/Q3W), pre-dose Week 9 (Q2W), pre-dose Week 10 (QW3) and pre-dose every 4 subsequent weeks and end of treatment (post-study: 4 weeks after last dose of study drug).
Time Frame: Up to 2 years
Population: The population consisted of all participants who received >90% of intended drug volume and had measurements at Baseline and at least once during treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dalotuzumab 1.25 mg/kg Q1W (10 mg/mL) | Dalotuzumab 2.5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (20 mg/mL) | Dalotuzumab 15 mg/kg Q1W (10 mg/mL) | Dalotuzumab 15 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q1W (10 mg/mL) | Dalotuzumab 20 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q2W (20 mg/mL) | Dalotuzumab 30 mg/kg Q3W (20 mg/mL)
Number analyzed (Participants) | 5 | 3 | 8 | 6 | 6 | 6 | 8 | 7 | 9 | 11 | 11
Percentage of Participants | 40 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 0 | 0 | 0

9. Secondary Outcome: Percentage of Participants Who Experienced a Complete Response (CR) or Partial Response (PR)
Description: Tumor responses were measured by using Response Evaluation Criteria in Solid Tumors (RECIST) criteria in participants with solid tumors and using European Group for Blood and Marrow Transplantation (EBMT) criteria in participants with multiple myeloma. RECIST criteria for CR: Disappearance of all target lesions. RECIST criteria for PR: ≥30% decrease in the sum of diameters of target lesions. EBMT criteria for CR: Disappearance of the original mAb protein from the blood and urine AND <5% plasma cells in the bone marrow AND no increase in the size or number of lytic bone lesions AND disappearance of soft tissue plasmacytomas AND normal serum calcium levels. EMBT criteria for PR: ≥50% reduction in the serum mAb protein level AND if a urine M-component is present, a reduction in 24-hour urinary light chain excretion by either ≥90% or to <200 mg AND ≥50% reduction in the size of soft tissue plasmacytomas AND no increase in size or number of lytic bone lesions.
Time Frame: Up to 2 years
Population: The population consisted of all evaluable participants who received >90% of intended drug volume and had efficacy measurements at Baseline and at least once during treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dalotuzumab 1.25 mg/kg Q1W (10 mg/mL) | Dalotuzumab 2.5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (20 mg/mL) | Dalotuzumab 15 mg/kg Q1W (10 mg/mL) | Dalotuzumab 15 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q1W (10 mg/mL) | Dalotuzumab 20 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q2W (20 mg/mL) | Dalotuzumab 30 mg/kg Q3W (20 mg/mL)
Number analyzed (Participants) | 5 | 3 | 8 | 6 | 6 | 6 | 8 | 7 | 9 | 11 | 11
Percentage of Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose of study drug (Up to 25 months)
Description: The population consisted of all participants who received at least one dose of study drug.
Groups:
- Dalotuzumab 15 mg/kg Q1W (20 mg/mL): Participants received dalotuzumab 15 mg/kg (20 mg/mL) IV infusion Q1W.
- Dalotuzumab 20 mg/kg Q1W (20 mg/mL): Participants received dalotuzumab 20 mg/kg (20 mg/mL) IV infusion Q1W.
Arm/Group | Dalotuzumab 1.25 mg/kg Q1W (10 mg/mL) | Dalotuzumab 2.5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 5 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (10 mg/mL) | Dalotuzumab 10 mg/kg Q1W (20 mg/mL) | Dalotuzumab 15 mg/kg Q1W (10 mg/mL) | Dalotuzumab 15 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q1W (10 mg/mL) | Dalotuzumab 20 mg/kg Q1W (20 mg/mL) | Dalotuzumab 20 mg/kg Q2W (20 mg/mL) | Dalotuzumab 30 mg/kg Q3W (20 mg/mL)
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3 | 2/8 | 2/6 | 2/6 | 3/6 | 3/8 | 0/7 | 2/9 | 3/11 | 1/11
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 6/8 | 5/6 | 4/6 | 5/6 | 8/8 | 6/7 | 8/9 | 9/11 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalotuzumab 1.25 mg/kg Q1W (10 mg/mL) (N=5) | Dalotuzumab 2.5 mg/kg Q1W (10 mg/mL) (N=3) | Dalotuzumab 5 mg/kg Q1W (10 mg/mL) (N=8) | Dalotuzumab 10 mg/kg Q1W (10 mg/mL) (N=6) | Dalotuzumab 10 mg/kg Q1W (20 mg/mL) (N=6) | Dalotuzumab 15 mg/kg Q1W (10 mg/mL) (N=6) | Dalotuzumab 15 mg/kg Q1W (20 mg/mL) (N=8) | Dalotuzumab 20 mg/kg Q1W (10 mg/mL) (N=7) | Dalotuzumab 20 mg/kg Q1W (20 mg/mL) (N=9) | Dalotuzumab 20 mg/kg Q2W (20 mg/mL) (N=11) | Dalotuzumab 30 mg/kg Q3W (20 mg/mL) (N=11)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ewing's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalotuzumab 1.25 mg/kg Q1W (10 mg/mL) (N=5) | Dalotuzumab 2.5 mg/kg Q1W (10 mg/mL) (N=3) | Dalotuzumab 5 mg/kg Q1W (10 mg/mL) (N=8) | Dalotuzumab 10 mg/kg Q1W (10 mg/mL) (N=6) | Dalotuzumab 10 mg/kg Q1W (20 mg/mL) (N=6) | Dalotuzumab 15 mg/kg Q1W (10 mg/mL) (N=6) | Dalotuzumab 15 mg/kg Q1W (20 mg/mL) (N=8) | Dalotuzumab 20 mg/kg Q1W (10 mg/mL) (N=7) | Dalotuzumab 20 mg/kg Q1W (20 mg/mL) (N=9) | Dalotuzumab 20 mg/kg Q2W (20 mg/mL) (N=11) | Dalotuzumab 30 mg/kg Q3W (20 mg/mL) (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 3 (5)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4)
Asthenia (General disorders) | 0 (0) | 2 (2) | 4 (5) | 2 (3) | 2 (2) | 0 (0) | 3 (5) | 2 (3) | 2 (2) | 3 (3) | 5 (6)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 3 (4) | 1 (2) | 1 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 2 (2) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 4 (5) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (4) | 1 (3) | 1 (1) | 3 (6) | 2 (3) | 1 (2) | 3 (4) | 1 (3) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (8) | 1 (1) | 2 (2) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (6) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.